CLINICAL TRIAL: NCT02320422
Title: An Intervention to Improve Adherence to Medications in Adults With Liver Transplants
Brief Title: Adult Liver Transplant Enhanced Care
Acronym: ALTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-1876
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Liver Transplant Recipients
Keywords: liver transplant; medication adherence; intervention
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral Telehealth (Experimental)
  Interventions: Behavioral: Behavioral Telehealth

INTERVENTIONS:
Behavioral: Behavioral Telehealth — The telemetric intervention (administered via telephone, or interactive video chat applications such as FaceTime ® or Skype ®) will enable the intervention team (IT) to address non-adherence from a remote location, using a structured, tailored approach

SUMMARY:
The purpose of this study is to pilot-test a tailored telemetric intervention to improve adherence to medications in adults who had a liver transplant and are presently non-adherent (as measured by tacrolimus levels).

DETAILED DESCRIPTION:
Adult patients who received a liver transplant and for whom there are at least 3 tacrolimus blood levels within the last year are eligible for the study. Patients will be recruited from amongst the roster of liver transplant recipients treated at the Recanati-Miller Transplant Institute at Mount Sinai. The intervention will be pilot-tested on up to 15 non-adherent patients. Patients will be identified using an innovative biomarker for non-adherence-by calculating the degree of fluctuation between individual medication blood levels. The telemetric intervention (administered via telephone, or interactive video chat applications such as FaceTime ® or Skype ®) will enable the intervention team (IT) to address non-adherence from a remote location, using a structured, tailored approach that accommodates specific patient needs. The approach includes a focus on psychological avoidance.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age.
* The patient received a liver transplant at least 2 years prior to initiation of the research protocol.
* The patient is able to provide consent (i.e. is not encephalopathic or does not have significant cognitive impairment). Consent may be obtained either by phone or in person (following a script) and is documented by the researcher.
* The patient is prescribed tacrolimus (either brand or generic formulation).
* The patient is not receiving Hepatitis C treatment during the intervention (given this can affect levels of tacrolimus and adherence behaviors)
* Thee patient has been seen in the liver transplant clinic at least once in the last two years.
* The patient's MLVI value was ≥ 2, with at least 3 levels present to make this determination. Only tacrolimus levels drawn in the outpatient setting will be included in SD calculations. Tacrolimus levels in the inpatient setting (i.e. during a hospitalization) will be excluded.
* The patient speaks English or Spanish at a level that allows him/her to understand the study procedures and consent to the study.

Exclusion Criteria:

* The patient received a liver transplant less than 2 years prior to enrollment.
* The patient received a dual transplant (i.e. liver and kidney).
* The treating physician has instructed the patient not to obtain tacrolimus levels for at least one year in the past year.
* The patient does not understand the study procedures. This will be verified by asking the patient to repeat the study procedures.
* The patient is actively psychotic or severely disoriented due to any cause, including hepatic encephalopathy (temporary exclusion) or severe cognitive impairment.
* The patient is not medically stable or is hospitalized (temporary exclusion until stabilized).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Medication Level Variability Index (MLVI) | up to 1 year
  The degree of fluctuation of tacrolimus blood levels (calculated as the standard deviation, SD, of tacrolimus).

SECONDARY OUTCOMES:
Incidence of biopsy-proven rejection | up to 1 year
  The number of incidences of liver transplant rejection (as proven by biopsy).
ALT | up to 1 year
  Liver enzyme levels - mean/maximum levels of ALT
Incidence of hospitalizations | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shemesh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States